CLINICAL TRIAL: NCT00865904
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Study of VX-809 to Evaluate Safety, Pharmacokinetics, and Pharmacodynamics of VX-809 in Cystic Fibrosis Subjects Homozygous for the ∆F508-CFTR Gene Mutation
Brief Title: Study of VX-809 in Cystic Fibrosis Subjects With the ∆F508-CFTR Gene Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VX08-809-101
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Results first posted 2015-08-28 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-06

CONDITIONS: Cystic Fibrosis
Keywords: ∆F508; F508del; Cystic Fibrosis Transmembrane Conductance Regulator; CFTR; Pancreatic diseases; Lung diseases; Genetic disease, inborn; Infant, newborn, diseases
MeSH Terms: conditions — Cystic Fibrosis; Pancreatic Diseases; Lung Diseases; Genetic Diseases, Inborn; Infant, Newborn, Diseases | interventions — lumacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Placebo matched to VX-809 capsule orally once daily for 28 days.
  Interventions: Drug: Placebo
- VX-809, 25 mg (Experimental): VX-809, 25 milligram (mg) capsule orally once daily for 28 days.
  Interventions: Drug: VX-809
- VX-809, 50 mg (Experimental): VX-809, 50 mg capsule orally once daily for 28 days.
  Interventions: Drug: VX-809
- VX-809, 100 mg (Experimental): VX-809, 100 mg capsule orally once daily for 28 days.
  Interventions: Drug: VX-809
- VX-809, 200 mg (Experimental): VX-809, 200 mg capsule orally once daily for 28 days.
  Interventions: Drug: VX-809

INTERVENTIONS:
Drug: VX-809 — Capsules
  Arms: VX-809, 100 mg; VX-809, 200 mg; VX-809, 25 mg; VX-809, 50 mg
Drug: Placebo — Placebo matched to VX-809 capsules.
  Arms: Placebo

SUMMARY:
The primary objective of the study was to evaluate the safety and tolerability of VX-809 in participants with cystic fibrosis (CF) who are homozygous for the F508del mutation on the CF transmembrane conductance regulator (CFTR) gene.

DETAILED DESCRIPTION:
This was a Phase 2, randomized, double-blind, placebo-controlled, multiple-dose study of orally-administered VX-809 in participants with CF who are homozygous for the specific CFTR mutation known as ∆F508 or F508del. Enrollment was planned for 90 participants at approximately 20 centers. Participants were planned to be randomized in a 4:1 ratio to receive 1 of 4 doses of VX-809 or placebo once a day for 28 days in a parallel design. Participants were outpatients during the study, except for overnight stays on Day 1 and 28.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF with ∆F508-CFTR mutation in both alleles
* Forced expiratory volume in 1 second (FEV1) greater than or equal to (>=) 40 percent (%) of predicted normal for age, gender, and height
* Weight >=40 kilograms (kg) and body mass index greater than or equal to 18.5 kilogram per square meter (kg/m^2)
* Screening laboratory values, tests, and physical examination within acceptable ranges
* Negative pregnancy test (for women of child-bearing potential)
* Able and willing to follow contraceptive requirements
* Willing to remain on a stable medication regimen for the duration of study participation

Exclusion Criteria:

* History of any illness, or any ongoing acute illness, that could impact the safety of the study participant or may confound results of study
* Pulmonary exacerbation or changes in therapy for pulmonary disease within 14 days before receiving the first dose of study drug
* Impaired hepatic or renal function
* History of organ or hematological transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (25):
- United States (18):
  - Birmingham, Alabama
  - Palo Alto, California
  - San Diego, California
  - Aurora, Colorado
  - Atlanta, Georgia
  - Chicago, Illinois
  - Iowa City, Iowa
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Seattle, Washington
- Belgium (2):
  - Brussels
  - Leuven
- Toronto, Ontario, Canada
- Germany (2):
  - Cologne
  - Hanover
- Netherlands (2):
  - Rotterdam
  - Utrecht

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662
- [Derived] Clancy JP, Rowe SM, Accurso FJ, Aitken ML, Amin RS, Ashlock MA, Ballmann M, Boyle MP, Bronsveld I, Campbell PW, De Boeck K, Donaldson SH, Dorkin HL, Dunitz JM, Durie PR, Jain M, Leonard A, McCoy KS, Moss RB, Pilewski JM, Rosenbluth DB, Rubenstein RC, Schechter MS, Botfield M, Ordonez CL, Spencer-Green GT, Vernillet L, Wisseh S, Yen K, Konstan MW. Results of a phase IIa study of VX-809, an investigational CFTR corrector compound, in subjects with cystic fibrosis homozygous for the F508del-CFTR mutation. Thorax. 2012 Jan;67(1):12-8. doi: 10.1136/thoraxjnl-2011-200393. Epub 2011 Aug 8. PMID 21825083

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | VX-809, 25 mg | VX-809, 50 mg | VX-809, 100 mg | VX-809, 200 mg
Started | 19 (Randomized.) | 18 (Randomized.) | 18 (Randomized.) | 18 (Randomized.) | 20 (Randomized.)
Completed | 17 (Completed 14-day follow-up.) | 18 (Completed 14-day follow-up.) | 18 (Completed 14-day follow-up.) | 17 (Completed 14-day follow-up.) | 19 (Completed 14-day follow-up.)
Not Completed | 2 | 0 | 0 | 1 | 1
Not completed — Randomized but not Treated | 2 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug.
Groups:
- VX-809, 25 mg: VX-809, 25 mg capsule orally once daily for 28 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | VX-809, 25 mg | VX-809, 50 mg | VX-809, 100 mg | VX-809, 200 mg | Total
Number analyzed (Participants) | 17 | 18 | 18 | 17 | 19 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (9.35) | 27.7 (8.98) | 27.1 (8.20) | 30.1 (11.55) | 26.7 (6.82) | 28.6 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 9 | 5 | 7 | 36
  Male | 11 | 9 | 9 | 12 | 12 | 53

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability Based on Adverse Events (AEs)
Description: AE: any untoward medical occurrence in a participant during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or previous condition that has increased in severity or frequency after the informed consent form is signed. AE includes serious as well as Non-serious AEs. Serious adverse event (SAE) (subset of AE): medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, in-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. Number of participants with AEs and SAEs are reported. An AE that started at or after initial dosing of study drug, or increased in severity after initial dosing of study drug visit is considered treatment-emergent.
Time Frame: Up to 14 days after last dose (last dose = Day 28)
Population: Safety set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | VX-809, 25 mg | VX-809, 50 mg | VX-809, 100 mg | VX-809, 200 mg
Number analyzed (Participants) | 17 | 18 | 18 | 17 | 19
participants
  Participants With Any AE | 17 | 16 | 15 | 16 | 18
  Participants With SAE | 1 | 5 | 1 | 0 | 3

2. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Day 28
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Baseline, Day 28
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug. Number of participants analyzed signifies participants evaluable for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: liters
Arm/Group | Placebo | VX-809, 25 mg | VX-809, 50 mg | VX-809, 100 mg | VX-809, 200 mg
Number analyzed (Participants) | 17 | 17 | 17 | 16 | 18
liters | 0.029 [-0.0823 to 0.1398] | -0.049 [-0.1578 to 0.0588] | -0.031 [-0.1401 to 0.0787] | 0.015 [-0.0972 to 0.1263] | -0.009 [-0.1146 to 0.0970]

3. Secondary Outcome: Change From Baseline in Percent Predicted FEV1 at Day 28
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Predicted FEV1 (for age, gender, and height) was calculated using the Knudson method.
Time Frame: Baseline, Day 28
Population: FAS. Number of participants analyzed signifies participants evaluable for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent predicted of FEV1
Arm/Group | Placebo | VX-809, 25 mg | VX-809, 50 mg | VX-809, 100 mg | VX-809, 200 mg
Number analyzed (Participants) | 17 | 17 | 17 | 16 | 18
Percent predicted of FEV1 | 0.285 [-2.8268 to 3.3973] | -1.637 [-4.6836 to 1.4089] | -0.375 [-3.4540 to 2.7046] | 0.168 [-2.9653 to 3.3011] | -0.165 [-3.1346 to 2.8044]

4. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at Day 28
Description: FVC is the volume of air that can be forcibly exhaled from the lungs after taking the deepest breath possible.
Time Frame: Baseline, Day 28
Population: FAS. Number of participants analyzed signifies participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | VX-809, 25 mg | VX-809, 50 mg | VX-809, 100 mg | VX-809, 200 mg
Number analyzed (Participants) | 17 | 17 | 17 | 16 | 18
liters | 0.085 (0.2857) | -0.055 (0.2331) | -0.020 (0.3494) | -0.004 (0.1916) | -0.023 (0.3668)

5. Secondary Outcome: Change From Baseline in Forced Expiratory Flow Over the Middle Half of the FVC (FEF25-75) at Day 28
Description: FEF25-75 is total volume of air exhaled from the lungs over the middle half of the FVC test, expressed as liters per second (L/sec).
Time Frame: Baseline, Day 28
Population: FAS. Number of participants analyzed signifies participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: liters per second (L/sec)
Arm/Group | Placebo | VX-809, 25 mg | VX-809, 50 mg | VX-809, 100 mg | VX-809, 200 mg
Number analyzed (Participants) | 17 | 17 | 17 | 16 | 18
liters per second (L/sec) | -0.030 (0.1730) | -0.011 (0.3231) | -0.029 (0.4373) | 0.045 (0.2702) | -0.052 (0.3558)

6. Secondary Outcome: Change From Baseline in Sweat Chloride at Day 28
Description: Sweat samples were collected using an approved Macroduct (Wescor) collection device. A volume of greater than or equal to (>=) 15 microliter was required for determination of sweat chloride.
Time Frame: Baseline, Day 28
Population: FAS. Number of participants analyzed signifies participants evaluable for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Arm/Group | Placebo | VX-809, 25 mg | VX-809, 50 mg | VX-809, 100 mg | VX-809, 200 mg
Number analyzed (Participants) | 16 | 16 | 16 | 15 | 16
millimole per liter (mmol/L) | 0.84 [-3.493 to 5.166] | 0.93 [-3.308 to 5.173] | -3.77 [-7.966 to 0.416] | -5.29 [-9.618 to -0.963] | -7.38 [-11.590 to -3.166]

7. Secondary Outcome: Change From Baseline in Nasal Potential Difference (NPD) of Zero Chloride Plus Isoproterenol Response at Day 28
Description: Nasal potential difference (NPD) provides a direct and sensitive evaluation of sodium and chloride transport in secretory epithelial cells via assessment of transepithelial bioelectric properties. NPD under conditions of zero chloride concentration perfusion solution in the presence of isoproterenol is reported.
  NPDs were performed according to Cystic Fibrosis Foundation Therapeutics Development Network (CFFT TDN) Standard Operating Procedure (SOP) 528.00 "Standardization of Measurement of Nasal Membrane Transepithelial Potential Difference (NPD) - electronic data capture (EDC) and Perfusion or Perfusion-Free Probe".
Time Frame: Baseline, Day 28
Population: FAS. Number of participants analyzed signifies participants evaluable for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: millivolts (mV)
Arm/Group | Placebo | VX-809, 25 mg | VX-809, 50 mg | VX-809, 100 mg | VX-809, 200 mg
Number analyzed (Participants) | 12 | 16 | 13 | 11 | 12
millivolts (mV) | -1.017 [-3.2979 to 1.2637] | 0.832 [-1.1302 to 2.7943] | 0.142 [-2.0369 to 2.3208] | 1.382 [-0.9853 to 3.7491] | 1.583 [-0.6952 to 3.8612]

8. Secondary Outcome: Change From Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Domain Scores at Day 28
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. CFQ-R domains include: Body, Digestion, Eat, Emotion, Health Perceptions, Physical, Respiratory, Role, Social, Treatment Burden, Vitality, and Weight. Individual domain score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: Baseline, Day 28
Population: FAS. Number of participants analyzed signifies participants evaluable for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | VX-809, 25 mg | VX-809, 50 mg | VX-809, 100 mg | VX-809, 200 mg
Number analyzed (Participants) | 17 | 17 | 17 | 16 | 18
units on a scale
  Body | -1.341 [-6.4183 to 3.7370] | -0.206 [-5.2276 to 4.8151] | -1.626 [-6.6796 to 3.4276] | 2.611 [-2.5525 to 7.7746] | 0.058 [-4.8954 to 5.0123]
  Digestion | 4.620 [-0.2530 to 9.4935] | 2.284 [-2.4928 to 7.0605] | -0.719 [-5.5599 to 4.1216] | 0.251 [-4.6794 to 5.1810] | 2.578 [-2.1027 to 7.2580]
  Eat | 2.110 [-3.9925 to 8.2128] | -3.662 [-9.6704 to 2.3463] | -7.269 [-13.3216 to -1.2161] | 3.242 [-3.0242 to 9.5087] | -2.576 [-8.4313 to 3.2793]
  Emotion | 4.859 [-0.4200 to 10.1372] | -3.222 [-8.4312 to 1.9866] | -1.358 [-6.5817 to 3.8666] | 3.489 [-1.9312 to 8.9087] | -2.624 [-7.7058 to 2.4585]
  Health Perceptions | 5.034 [-1.6041 to 11.6713] | -2.839 [-9.2912 to 3.6131] | -6.967 [-13.4203 to -0.5137] | -0.435 [-7.0778 to 6.2074] | -1.896 [-8.3524 to 4.5604]
  Physical | 1.225 [-5.3271 to 7.7764] | -5.968 [-12.3586 to 0.4217] | -7.384 [-13.8167 to -0.9508] | -3.464 [-10.0613 to 3.1335] | -0.976 [-7.2596 to 5.3067]
  Respiratory | 4.534 [-1.6158 to 10.6842] | -5.223 [-11.2414 to 0.7956] | -6.324 [-12.3453 to -0.3026] | -1.290 [-7.5407 to 4.9598] | 2.215 [-3.6610 to 8.0901]
  Role | 2.210 [-3.2279 to 7.6481] | -5.941 [-11.3247 to -0.5577] | -4.599 [-9.9912 to 0.7925] | 1.097 [-4.4579 to 6.6510] | -6.533 [-11.7858 to -1.2803]
  Social | -0.554 [-4.8235 to 3.7152] | -0.001 [-4.2221 to 4.2200] | -1.013 [-5.2372 to 3.2122] | 0.469 [-3.8898 to 4.8273] | -2.640 [-6.7802 to 1.5008]
  Treatment Burden | 2.463 [-3.1916 to 8.1169] | 4.185 [-1.4220 to 9.7914] | -5.962 [-11.5712 to -0.3530] | 1.421 [-4.3528 to 7.1954] | -0.676 [-6.1363 to 4.7843]
  Vitality | -2.178 [-8.8193 to 4.4629] | -4.645 [-11.1048 to 1.8139] | -7.227 [-13.6961 to -0.7589] | -1.516 [-8.1800 to 5.1472] | 0.730 [-5.5932 to 7.0522]
  Weight | 0.304 [-9.4460 to 10.0543] | 5.410 [-4.2393 to 15.0600] | 2.175 [-7.5500 to 11.8997] | 8.827 [-1.1524 to 18.8063] | -4.186 [-13.5956 to 5.2233]

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) of VX-809
Description: Only participants who received VX-809 were analyzed for this outcome measure.
Time Frame: Day 1 (pre dose, 0.75, 1.5, 3, 4, 6, 9, 12, and 24 hours post-dose), Day 28 (pre dose, 0.75, 1.5, 3, 4, 6, 9, 12, 24, and 30-60 hours post dose)
Population: FAS. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | VX-809, 25 mg | VX-809, 50 mg | VX-809, 100 mg | VX-809, 200 mg
Number analyzed (Participants) | 18 | 18 | 17 | 19
nanogram per milliliter (ng/mL)
  Day 1 (n= 18, 18, 17, 19) | 760 (280) | 1850 (697) | 2930 (916) | 6410 (2550)
  Day 28 (n= 17, 17, 16, 18) | 1100 (443) | 2660 (1010) | 4620 (1840) | 10300 (4490)

10. Secondary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to 24 Hours (AUC0-24) of VX-809
Description: Only participants who received VX-809 were analyzed for this outcome measure.
Time Frame: Day 1 (pre dose, 0.75, 1.5, 3, 4, 6, 9, 12, and 24 hours post-dose), Day 28 (pre dose, 0.75, 1.5, 3, 4, 6, 9, 12, and 24 hours post dose)
Population: FAS. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | VX-809, 25 mg | VX-809, 50 mg | VX-809, 100 mg | VX-809, 200 mg
Number analyzed (Participants) | 18 | 18 | 17 | 19
hour*nanogram per milliliter (hr*ng/mL)
  Day 1 (n= 18, 18, 17, 19) | 7190 (2190) | 16600 (6290) | 29000 (11400) | 59500 (26400)
  Day 28 (n= 17, 17, 16, 18) | 12900 (4920) | 28800 (13100) | 54100 (31600) | 119000 (73700)

ADVERSE EVENTS:
Time Frame: Up to 14 days after last dose (last dose = Day 28)
Arm/Group | Placebo | VX-809, 25 mg | VX-809, 50 mg | VX-809, 100 mg | VX-809, 200 mg
Serious Adverse Events (participants affected / at risk) | 1/17 | 5/18 | 1/18 | 0/17 | 3/19
Other Adverse Events (participants affected / at risk) | 17/17 | 16/18 | 15/18 | 16/17 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=17) | VX-809, 25 mg (N=18) | VX-809, 50 mg (N=18) | VX-809, 100 mg (N=17) | VX-809, 200 mg (N=19)
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 1 | 4 | 1 | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=17) | VX-809, 25 mg (N=18) | VX-809, 50 mg (N=18) | VX-809, 100 mg (N=17) | VX-809, 200 mg (N=19)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 10 | 6 | 7 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 3 | 2 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 4 | 6
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 2 | 3 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 2 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 0 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0 | 1
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Lung hyperinflation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Nasal turbinate abnormality (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 1
Post-tussive vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Infrequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 3 | 3 | 2 | 3
Pyrexia (General disorders) | 2 | 2 | 1 | 1 | 5
Pain (General disorders) | 1 | 1 | 1 | 0 | 1
Chest discomfort (General disorders) | 1 | 1 | 0 | 0 | 0
Catheter site haematoma (General disorders) | 0 | 0 | 1 | 0 | 0
Catheter site rash (General disorders) | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0
Hunger (General disorders) | 0 | 0 | 0 | 0 | 1
Irritability (General disorders) | 0 | 0 | 0 | 1 | 0
Nodule (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
Breath sounds abnormal (Investigations) | 1 | 1 | 0 | 1 | 1
Forced expiratory volume decreased (Investigations) | 0 | 1 | 1 | 1 | 1
Pulmonary function test decreased (Investigations) | 1 | 1 | 0 | 1 | 1
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 2 | 0
Prothrombin time prolonged (Investigations) | 1 | 1 | 0 | 1 | 0
Sputum abnormal (Investigations) | 0 | 2 | 0 | 0 | 1
Blood glucose increased (Investigations) | 1 | 0 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 1 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0 | 0
Glucose urine (Investigations) | 0 | 0 | 1 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 1 | 0 | 0
Urine leukocyte esterase positive (Investigations) | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 4 | 5 | 2 | 5
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 2 | 1
Tension headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Sinus headache (Investigations) | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Clubbing (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1 | 3 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 2
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 1 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 1 | 1 | 1 | 2 | 1
Cystic fibrosis related diabetes (Congenital, familial and genetic disorders) | 1 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 1
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.